CLINICAL TRIAL: NCT06224101
Title: Heart-SIMS1: Simulation Training For Invasive Cardiovascular Procedures
Brief Title: Simulation Training For Invasive Cardiovascular Procedures
Acronym: Heart-SIMS1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Manuel Oliveira Santos, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Heart-SIMS1
Record Dates: First submitted 2024-01-14; First posted 2024-01-25 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Disease
Keywords: Education; Invasive coronary angiography; Cardiovascular procedures; 3D-printing; Simulation training
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional training group (No Intervention): The conventional training group will visualize a video-recorded simulation procedure with duration of 20 minutes, in which the steps of the ICA are explained.
- Simulation training group (Experimental): The simulation training group will perform coronary angiography simulated training with 3D printed simulator SimulHeart in groups of two, with debriefing and feedback. Participants will be taught on how to perform each step of the procedure and guide on safety measures concerning catheter handling, radiation exposure, and contrast administration. The duration of simulated training will be 20 minutes per group.
  Interventions: Behavioral: Simulation-based training

INTERVENTIONS:
Behavioral: Simulation-based training — simulation training consists of practicing diagnostic coronary angiography with 3D printed simulator-SimulHeart.
  Arms: Simulation training group

SUMMARY:
28 sixth-year medical students will attend a theoretical learning session on coronary angiography. After they will be randomized in 2 groups: a conventional training (CT) group (n=14) and a simulation training (ST) group (n=14). CT group will visualize a video-recorded simulation procedure with duration of 20 minutes, while ST group will perform CA simulated training with SimulHeart in groups of two also for 20 minutes. Finally, after the training session, students' knowledge will be assessed through a theoretical multiple-choice exam and a practical evaluation in a catheterization laboratory using SimulHeart.

DETAILED DESCRIPTION:
The simulation protocol starts with a theoretical learning session on invasive coronary angiography (ICA) (1 hour), encompassing the learning objectives (coronary anatomy, procedural indications and safety considerations) for all participants. During the theoretical session, students will be instructed on the most utilized tools for conducting coronary catheterization, along with a step-by-step sequence of the procedure. Medical students will be then randomized to two training methodologies (1:1) using Python programming language, at the same location: a conventional training (CT) group (n=14) and a simulation training (ST) group (n=14). No pre-testing will be performed, because medical students, unlike residents, have limited knowledge on ICA, and randomization will naturally balance both groups. The CT group will visualize a video-recorded simulation procedure with duration of 20 minutes, in which the steps of the ICA are explained. The ST group will perform ICA simulated training with 3D printed simulator SimulHeart in groups of two, with debriefing and feedback. Participants will be taught on how to perform each step of the procedure and guide on safety measures concerning catheter handling, radiation exposure, and contrast administration. The duration of ICA simulated training will be 20 minutes per group. Both types of sessions will have the same instructions and duration (20 minutes). There will be time for questions and answers. After the training session, students' knowledge will be assessed through a theoretical multiple-choice exam, assessing basic coronary artery anatomy knowledge, procedural indications, and safety considerations (scored 0-100 points) and a practical evaluation. The practical evaluation will take place in a catheterization laboratory using SimulHeart simulator at "Unidade de Intervenção Cardiovascular (UNIC), Serviço de Cardiologia do Centro Hospitalar e Universitário de Coimbra (Coimbra, Portugal)". The participants will have to perform pre-specified steps during practical session of diagnostic ICA. The procedure will be video-taped and rated based on performance time, execution of pre-specified steps and monitoring of safety requirements. The student's performance will be evaluated (scored 0-100 points) in real-time and subsequently through review and the analysis of the recorded videos by experts interventionalists, blinded to the randomization and under a checklist of pre-specified safety endpoints and a performance evaluation checklist.

ELIGIBILITY:
Inclusion Criteria:

* 6th-year medical students who have read and signed the informed consent

Exclusion Criteria:

* Pregnant students
* Previous experience in interventional cardiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-06-09 (Actual)

PRIMARY OUTCOMES:
Score of theoretical multiple-choice exam | 2 days
  Students' knowledge of both groups will be assessed through a theoretical multiple-choice exam, assessing basic coronary artery anatomy knowledge, procedural indications, and safety considerations (scored 0-100 points)
Score of pratical evaluation of simulated coronary angiography in a catheterization laboratory | 2 days
  Students' knowledge of both groups will be assessed through a practical evaluation in a catheterization laboratory using 3D-simulator SimulHeart. The students will have to performe pre-specified steps during pratical session (scored 0-100 points)
Final performance score (0-200 points) | 2 days
  Composite endpoint resulting from the sum of the practical evaluation score and the multiple-choice theoretical test score

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Oliveira Santos, MD, Principal Investigator — Coimbra's University - Faculty of Medicine
Locations (1):
- Centro Hospitalar e Universitário de Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fischer Q, Sbissa Y, Nhan P, Adjedj J, Picard F, Mignon A, Varenne O. Use of Simulator-Based Teaching to Improve Medical Students' Knowledge and Competencies: Randomized Controlled Trial. J Med Internet Res. 2018 Sep 24;20(9):e261. doi: 10.2196/jmir.9634. PMID 30249587
- [Background] Popovic B, Pinelli S, Albuisson E, Metzdorf PA, Mourer B, Tran N, Camenzind E. The Simulation Training in Coronary Angiography and Its Impact on Real Life Conduct in the Catheterization Laboratory. Am J Cardiol. 2019 Apr 15;123(8):1208-1213. doi: 10.1016/j.amjcard.2019.01.032. Epub 2019 Jan 24. PMID 30732853
- [Background] Prenner SB, Wayne DB, Sweis RN, Cohen ER, Feinglass JM, Schimmel DR. Simulation-based education leads to decreased use of fluoroscopy in diagnostic coronary angiography. Catheter Cardiovasc Interv. 2018 May 1;91(6):1054-1059. doi: 10.1002/ccd.27203. Epub 2017 Aug 2. PMID 28766876
- [Background] Oliveira-Santos M, Oliveira Santos E, Marinho AV, Leite L, Guardado J, Matos V, Pego GM, Marques JS. Patient-specific 3D printing simulation to guide complex coronary intervention. Rev Port Cardiol (Engl Ed). 2018 Jun;37(6):541.e1-541.e4. doi: 10.1016/j.repc.2018.02.007. Epub 2018 May 7. English, Portuguese. PMID 29748151
- [Background] Voelker W, Petri N, Tonissen C, Stork S, Birkemeyer R, Kaiser E, Oberhoff M. Does Simulation-Based Training Improve Procedural Skills of Beginners in Interventional Cardiology?--A Stratified Randomized Study. J Interv Cardiol. 2016 Feb;29(1):75-82. doi: 10.1111/joic.12257. Epub 2015 Dec 16. PMID 26671629